CLINICAL TRIAL: NCT04829929
Title: Prospective, Single-arm Study to Assess the Safety and Performance of the Omega™ Left Atrial Appendage (LAA) Occluder in Patients With Non-Valvular Atrial Fibrillation and High Bleeding Risk
Brief Title: Evaluation of Safety and Performance of the Omega™ LAA (Left Atrial Appendage) Occluder and Omega™ Delivery System in Patients With Non-Valvular Atrial Fibrillation and High Bleeding Risk
Acronym: Omega
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eclipse Medical Ltd. (Industry)
Collaborators: KCRI (Other); Cardiovascular Research Institute Dublin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Omega
Record Dates: First submitted 2021-03-24; First posted 2021-04-02 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Non-Valvular Atrial Fibrillation
Keywords: non-valvular atrial fibrillation; left atrial appendage; occluder; LAA occluder; high bleeding risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm (Experimental): Patients with Non-Valvular Atrial Fibrillation and High Bleeding Risk
  Interventions: Device: Omega™LAA Occluder implantation

INTERVENTIONS:
Device: Omega™LAA Occluder implantation — Left Atrial Appendage closure for patients with non-valvular atrial fibrillation (NVAF) and high bleeding risk by Omega™LAA Occluder using Omega™ Delivery System

SUMMARY:
The purpose of the study is to assess the safety and performance of the Omega™ LAA (Left Atrial Appendage) Occluder and Omega™ Delivery System in LAA (Left Atrial Appendage) closure for patients with non-valvular atrial fibrillation (NVAF) and high bleeding risk.

DETAILED DESCRIPTION:
Omega™ LAA (Left Atrial Appendage) Occluder used in combination with the indicated Omega™ Delivery System is a permanent implant to the left atrial appendage for percutaneous insertion. LLA (Left Atrial Appendage) occlusion appears to be a feasible option for stroke reduction in AF patients at high risk for stroke, who are contraindicated for anticoagulation or who suffered a stroke despite OC. This study will evaluate safety and performance, using a study design which is based on inputs from pre-clinical testing, the risk analysis and data available from other LAA (Left Atrial Appendage) devices.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Documented paroxysmal, persistent, or permanent non-valvular atrial fibrillation (AF)
3. At increased risk of stroke or systemic embolism defined as a CHA2DS2-VASc score > or = 2
4. To have suitable anatomy for percutaneous Left Atrial Appendage occlusion procedure with a single Omega™ device
5. Able and willing to comply with the required medication regimen post-device implant
6. Able to understand and willing to provide written informed consent to participate in the study

Exclusion Criteria:

1. Requires long-term oral anticoagulation therapy for any indication other than atrial fibrillation
2. Contraindicated for or allergic to aspirin, clopidogrel, warfarin or novel oral anticoagulant (NOAC) use
3. Has any contraindications for a percutaneous catheterization procedure (e.g. subject is too small to accommodate the transoesophageal echocardiogram (TEE/TOE) probe or required catheters, or subject has active infection or bleeding disorder)
4. Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment per physician discretion)
5. Stroke or transient ischemic attack (TIA) within 6 weeks prior to implant procedure
6. Myocardial infarction (MI) within 90 days prior to implant
7. New York Heart Association Class IV Congestive Heart Failure
8. Left ventricular ejection Fraction (LVEF) < or = 30%
9. Left atrial appendage is obliterated or surgically ligated
10. Actively enrolled or plans to enrol in a concurrent clinical study in which the active treatment arm may confound the results of this trial
11. Active endocarditis or other infection producing bacteraemia
12. Subject has a known malignancy or other illness where life expectancy is less than 2 years
13. Impaired renal function with eGFR <30 ml/min/1.73 m2

Echocardiographic Exclusion Criteria:

1. Intracardiac thrombus - including LAA - visualized by echocardiographic imaging
2. Significant mitral valve stenosis (i.e. mitral valve area <1.5 cm2)
3. Cardiac tumour
4. LAA anatomy cannot accommodate an Omega™ device (as per IFU)
5. Placement of the device would interfere with any intracardiac or intravascular structure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
LAA (Left Atrial Appendage) closure | According to the local standards of care post-procedural, up to 3 months (First in-hospital follow-up visit which will take place after the procedure - depending on local treatment standards).
  The LAA closure is defined as complete seal or efficient seal with a peri-device leak ≤ 5 mm and assessed by Transthoracic or Transoesophageal Echo or cardiac computed tomography, with colour flow Doppler.
Device related complications | According to the local standards of care post-procedural, up to 3 months (First in-hospital follow-up visit which will take place around after the procedure - depending on local treatment standards).
  Serious adverse events (SAE)

SECONDARY OUTCOMES:
Procedure-related complications | Up to 7 days post-procedure
  All Serious Adverse Events
Device-related complications | 24 months
  All Serious Adverse Events including device thrombus
Major bleeding | 24 months
  Major bleeding defined as ≥ BARC (Bleeding Academic Research Consortium) 3 bleed
Ischemic stroke | 24 months
  Confirmed by Neurologic assessment and appropriate CT (Computed Tomography)/MR (Magnetic Resonance) imaging
Systemic embolism | 24 months
  Confirmed by appropriate imaging
Pericardial effusion/tamponade | 24 months
  Confirmed by appropriate imaging
Technical success at implant | According to the local standards of care post-procedural, up to 3 months (First in-hospital follow-up visit which will take place around after the procedure - depending on local treatment standards).
  No device-related complications, occlusion of the left atrial appendage
Procedural success | According to the local standards of care post-procedural, up to 3 months (First in-hospital follow-up visit which will take place around after the procedure - depending on local treatment standards).
  Technical success, no procedure-related complications except uncomplicated (minor) device embolization resolved by percutaneous retrieval during the procedure without surgical intervention or damage to surrounding cardiovascular structures

CONTACTS AND LOCATIONS:
Overall Officials: Horst Sievert, profesor, Principal Investigator — Cardio Vasculares Centrum, Seckbacher Landstrasse 65, 60389 Frankfurt, Germany
Locations (13):
- Denmark (2):
  - Rigshospitalet, Kardiologisk klinik B 2011, Copenhagen, Blegdamsvej 9
  - Aarhus University Hospital, Aarhus
- Germany (4):
  - CardioVasculäres Centrum, Seckbacher Landstrasse 65, Frankfurt, Frankfurt
  - Charité - University Medicine Berlin - Campus Benjamin Franklin, Berlin, Hindenburgdamm 30
  - Herzzentrum Leipzig, Leipzig, Strümpellstraße 39
  - Cardioangiologisches Centrum Bethanien, Frankfurt, Wilhelm-Epstein-Str. 4
- Mater Private Network, Dublin, Ireland
- Università Campus Biomedico Roma, Rome, Via Álvaro Del Portillo, 200, Italy
- Spain (4):
  - Instituto de Ciencias del Corazón (ICICOR) . Hospital Clínico Universitario, Valladolid, Avda. Ramón Y Cajal 3
  - Hospital Clinico San Carlos, Madrid, Calle Del Prof Martín Lagos
  - Complejo Hospitalario de Salamanca, Salamanca, Junta de Castilla Y LeónPaseo de San Vicente
  - Hospital de la Santa Creu I Sant Pau, Barcelona, Sant Antoni Maria Clare
- University Hospitals Sussex NHS Foundation Trust Clinical Research Facility, Brighton, East Sussex, United Kingdom

REFERENCES:
- [Background] De Backer O, Hafiz H, Fabre A, Lertsapcharoen P, Srimahachota S, Foley D, Sondergaard L. State-of-the-art preclinical testing of the OMEGATM left atrial appendage occluder. Catheter Cardiovasc Interv. 2021 Jun 1;97(7):E1011-E1018. doi: 10.1002/ccd.29331. Epub 2020 Oct 9. PMID 33034944